CLINICAL TRIAL: NCT04024670
Title: The Impact of Arts-Based Interventions on Patient Hospital Experience for Patients on a High-Risk Obstetrics and Bone Transplant Units
Brief Title: The Impact of Arts-Based Interventions on Patient Hospital Experience
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Kimberly Kirklin, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB-300001347; UL 1 TR003096 (Other: UAB)
Record Dates: First submitted 2019-04-25; First posted 2019-07-18 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: High Risk Pregnancy; Bone Marrow
Keywords: arts in medicine; sewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Patients on a high-risk obstetrics unit with an anticipated stay of two or more weeks (Active Comparator): patients in this group will receive twice weekly sewing and embroidery interactions with a professional artist in residence.
  Interventions: Other: Arts Intervention
- Patients on a bone marrow transplant unit with an anticipated stay of two or more weeks (Active Comparator): patients in this group will receive twice weekly visits with a professional storyteller.
  Interventions: Other: Arts Intervention
- HRO Standard of Care (No Intervention): SOC
- BMT Standard of Care (No Intervention): SOC

INTERVENTIONS:
Other: Arts Intervention — If selected for the arts activity, an artist in residence will visit you 3 times a week for a total of 3 weeks during your hospital stay. Two visits will focus on the arts activity and one visit will be the administration of the questionnaire. Each visit will be approximately 25 minutes at a time.
  Arms: Patients on a bone marrow transplant unit with an anticipated stay of two or more weeks; Patients on a high-risk obstetrics unit with an anticipated stay of two or more weeks

SUMMARY:
nuts and bolts

DETAILED DESCRIPTION:
interventions and timing of interventions

ELIGIBILITY:
Inclusion:

* Inpatient on either Bone Marrow Transplant ICU or High Risk Obstetrics Unit
* Estimated length of stay 2 or more weeks
* Age >18
* Patients who will potentially benefit from the AIM experience

Additional Inclusion Criteria:

* For the High Risk Obstetrics Unit group (hand-sewing), patients should be physically able to participate in hand-sewing activity.
* For the Bone Marrow Transplant IUC group (story-telling/poetry), patients should be physically able to participate in story-telling/poetry activity.

Exclusion:

* Patient too ill
* Complex medical condition that requires therapies which would not allow time for participation
* Declined to participate
* Age <18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Evaluate patient experience during the course of intervention using name of survey | Baseline at admissions
  define survey - evaluate experiences, range of survey - explain likert scale 0-10 with 0 being x (allows patient to rate how much they disagree or agree with a statement), 0 being the worst outcome and 10 being the best
Evaluate patient experience during the course of intervention using name of survey | Baseline - end of week 1
  define survey - evaluate experiences, range of survey - explain likert scale 0-10 with 0 being x (allows patient to rate how much they disagree or agree with a statement), 0 being the worst outcome and 10 being the best
Evaluate patient experience during the course of intervention using name of survey | week 1- week 2
  define survey - evaluate experiences, range of survey - explain likert scale 0-10 with 0 being x (allows patient to rate how much they disagree or agree with a statement), 0 being the worst outcome and 10 being the best
Evaluate patient experience during the course of intervention using name of survey | week 2 - week 3
  define survey - evaluate experiences, range of survey - explain likert scale 0-10 with 0 being x (allows patient to rate how much they disagree or agree with a statement), 0 being the worst outcome and 10 being the best
Evaluate patient experience during the course of intervention using name of survey | week 3 - weekly up to 10 weeks
  define survey - evaluate experiences, range of survey - explain likert scale 0-10 with 0 being x (allows patient to rate how much they disagree or agree with a statement), 0 being the worst outcome and 10 being the best

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly P Kirklin, MA, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
At this time we do not have IRB approval to share IPD. We may change this in the future.